CLINICAL TRIAL: NCT04664907
Title: Phenomenological Crossing of the Psychic Trauma and Its Resolution. Imagination at the Heart of the Treatment: Video-music as a Metaphor for Psychological Trauma and Its Resolution.
Brief Title: Videomusic and Psychic Trauma
Acronym: VIMUTRAU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Denied by Human Subjects Protection Board
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-CHITS-07; 2020-A02649-30 (Other: Id-RCB)
Record Dates: First submitted 2020-11-25; First posted 2020-12-11 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Psychic trauma; Phenomenology; Consciousness; Anxiety; Music; Videomusic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients suffering from post traumatic stress disorder (Experimental)
  Interventions: Other: Videomusic listening

INTERVENTIONS:
Other: Videomusic listening — Patients will attend a 8 min videomusic session and questionnaires will be performed before and after this session.

SUMMARY:
This project is interested in the flow of consciousness and its modalizations during psychological trauma (post-traumatic stress disorder) and its resolution. It is based on the premise that in PTSD, consciousness becomes more rigid, less fluid, due to the memory always imposing itself on the consciousness. The resolution of the trauma and the subsequent reduction of anxiety might improve the fluidity of consciousness and thus lead to an overall improvement in the psychological state of PTSD patients. In cases of PTSD, music has been shown to reduce anxiety from the very first session and has a very positive effect on all PTSD symptoms.

In this project the following elements will be evaluated : on one hand, the changes in consciousness and its fluidity and, on the other hand, the evolution of anxiety following the listening of a new kind of work, videomusic (which associates a video scenario with music) exemplifying (metaphorizing) the trauma and its resolution.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* Patients diagnosed with Simple Post Traumatic Stress according to DSM 5 criteria
* Patient able to express consent prior to participation in the study
* Patient affiliated to or beneficiary of a social security regimen

Exclusion Criteria:

* Other serious psychiatric pathologies
* Serious chronic pathologies, especially neurological ones
* Epilepsy
* Blindness or deafness
* Psychiatric decompensation
* Pregnant Women
* Patient under judicial protection (guardianship, curatorship...) or justice safeguard
* Any other reason that, in the opinion of the investigator, could interfere with study objective evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Consciousness fluidity using a questionnaire dedicated to this measure | 4 weeks
  Consciousness fluidity will be assessed before and after videomusic listening from the scores obtained at a questionnaire Evaluating Qualitatively the Fluidity of Consciousness (EQFC). Minimum and maximum values are 1 for "Never" and 6 for "Always". For some items, 1 indicates a better outcome and for some it is the contrary.

SECONDARY OUTCOMES:
Qualitative analysis of experiential phenomenological interview | 4 weeks
  Experiential phenomenological interview will be analyzed according to qualitative analyze criteria (occurrence frequencies)
Salience-resonances method | 4 weeks
  Experiential phenomenological interview will be analyzed according to salience-resonance method
Patient anxiety | 4 weeks
  Patient anxiety level will be analyzed before and after videomusic listening thanks to State-Trait Anxiety Inventory (STAI) scale and scores obtained will be correlated with EQFC scores. For each item scores go from 1 to 4. For some of them 1 means "Not at all" and 4 "A lot" and for others it is the contrary. A global score superior to 65 indicates a high level of anxiety and a global score inferior or equal to 35 a very low level of anxiety.
Post traumatic stress disorder phenomenological definition | 4 weeks
  Principal component analysis will be performed to find potential correlations between population initial characteristics and improvement of consciousness fluidity after videomusic listening

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Dias Alves, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer

IPD SHARING:
Plan to Share IPD: No